CLINICAL TRIAL: NCT01335620
Title: An Open Label Study to Investigate the Safety, Pharmacokinetic Profile and Efficacy of Raltegravir in HIV-infected Patients at Least 60 Years of Age
Brief Title: The Safety, Pharmacokinetic Profile and Efficacy of Raltegravir in HIV-infected Patients at Least 60 Years of Age
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTG_60; 2010-022907-23 (EudraCT Number)
Record Dates: First submitted 2011-03-25; First posted 2011-04-14 (Estimated); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: HIV
Keywords: HIV; Pharmatokinetic; 60 years old; Raltegravir
MeSH Terms: interventions — Raltegravir Potassium; Tenofovir; Emtricitabine

STUDY DESIGN:
Intervention Model Description: HIV affected over 60 years old
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tenofovir/Emtricitabine and Raltegravir (Other): Single arm study
  tenofovir/emtricitabine 245/200 mg once daily and raltegravir 400 mg twice daily
  Interventions: Drug: Raltegravir; Drug: Tenofovir; Drug: Emtricitabine

INTERVENTIONS:
Drug: Raltegravir — 400 mg twice daily
  Other Names: Isentress
Drug: Tenofovir — 245 mg once daily
Drug: Emtricitabine — 200mg once daily

SUMMARY:
This is a phase IV, open label, prospective, one phase pharmacokinetic and observational study.

Twenty HIV-1 infected subjects will be recruited, subjects will switch antiretroviral therapy to:

* tenofovir/emtricitabine 245/200 mg daily (Truvada™) plus
* raltegravir 400 mg twice daily On day 28, all subjects will attend for an intensive 24 hour pharmacokinetic visit.

DETAILED DESCRIPTION:
This is a phase IV, open label, prospective, one phase pharmacokinetic and observational study.

Twenty HIV-1 infected subjects will be recruited. Eligible subjects will currently be receiving stable antiretroviral therapy with undetectable plasma HIV RNA and have no evidence of previous HIV- resistance mutations on genotypic resistance testing.

At baseline, subjects will switch antiretroviral therapy to:

* tenofovir/emtricitabine 245/200 mg daily (Truvada™) plus
* raltegravir 400 mg twice daily On day 28, all subjects will attend for an intensive 24 hour pharmacokinetic visit.

Follow up over 6 months, subjects will attend on days 14, 90 and 180 for follow up visits that will include standard safety parameters. Assessment of cardiac biomarkers at baseline and on days 90 and 180 and assessment of neurocognitive function at screening, baseline and on day 180 will also be undertaken.

Following completion of this study, subjects will recommence their usual antiretroviral treatment regimen and attend for a study follow up visit.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected males or females
2. 60 years of age or greater*
3. signed informed consent
4. willing to switch therapy as per study protocol
5. no previous exposure to raltegravir or HIV-1 integrase inhibitors
6. plasma HIV RNA < 50 copies/mL at screening and on at least one other occasion over the last 3 months
7. currently receiving a stable antiretroviral regimen with no antiretroviral drug switches for at least 3 months
8. no previous clinically-significant resistance documented on HIV-1 genotypic resistance
9. subjects in good health upon medical history, physical exam, and laboratory testing
10. BMI above or equal to 18 and below 32
11. Male subjects who are heterosexually active must use two forms of barrier contraception (e.g., condom with spermicide) during heterosexual intercourse, from screening through completion of the study.
12. Have local screening laboratory results (haematology and chemistry that fall within the normal range of the central laboratory's reference ranges unless the results have been determined by the Investigator to have no clinical significance * 50% of total enrolled cohort will be 65 years of age or over. Subsequent to 10 subjects aged between 60 and 64 recruited, only subjects aged 65 or over will be eligible.

Exclusion Criteria:

1. current alcohol abuse or drug dependence
2. positive urine drug of abuse screening
3. active opportunistic infection or significant co-morbidities
4. current disallowed concomitant medication

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Winston, MB BH, Principal Investigator — Imperial College London; Marta Boffito, Principal Investigator — Chelsea & Westminster Hospital
Locations (2):
- United Kingdom (2):
  - Chelsea & Westminster Hospital NHS Trust, London
  - Imperial College Healthcare NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vera JH, Jackson A, Dickinson L, Else L, Barber T, Mora-Peris B, Back D, Boffito M, Winston A. The pharmacokinetic profile of raltegravir-containing antiretroviral therapy in HIV-infected individuals over 60 years of age. HIV Clin Trials. 2015 Jan-Feb;16(1):39-42. doi: 10.1179/1528433614Z.0000000006. Epub 2015 Jan 14. PMID 25777188

RESULTS

PARTICIPANT FLOW:
Groups:
- Truvada Plus Raltegravir: Single arm study
  Raltegravir: 400 mg twice daily
Period: Overall Study
Arm/Group | Truvada Plus Raltegravir
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Truvada Plus Raltegravir
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 19

OUTCOME MEASURES:

1. Primary Outcome: Drug Levels in Blood
Description: rategravir concentration
Time Frame: Day 28
Measure: Geometric Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Truvada Plus Raltegravir
Number analyzed (Participants) | 19
ng/ml | 1732 [969 to 3095]

2. Primary Outcome: Changes in Haematology, Biochemistry and Virology Tests
Description: full blood count, electrolytes and blood lipids will be measured at all visits to assess for changes through out the study. HIV viral load will also be measured to assess the efficacy of the medication at controlling the virus
Time Frame: 6 months
Population: No data collected
Arm/Group | Truvada Plus Raltegravir
Number analyzed (Participants) | 0

3. Secondary Outcome: Cardiovascular Disease Markers
Description: • To investigate cardiovascular disease markers before and after a switch in antiretroviral therapy to raltegravir.
Time Frame: 6 months
Population: No data collected
Arm/Group | Truvada Plus Raltegravir
Number analyzed (Participants) | 0

4. Secondary Outcome: Cerebral Function; Changes in Global Cognitive Z-score
Description: Cerebral function via cognitive testing before and after a switch in antiretroviral therapy to raltegravir.
  Mean Scores from the eight tasks (NPZ-8) assessed were used to derive a global composite measure of neurocognitive function. The result shows the change before and after switch, an increase in z-score represents an improvement in cognitive function assessed by CogState battery, required approximately 10-15 min for completion.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Truvada Plus Raltegravir
Number analyzed (Participants) | 19
score on a scale | 0.91 (1.3)
Statistical Analysis 1: Comparison: Truvada Plus Raltegravir; Compare baseline to 24 weeks; Test type: Superiority; p = 0.018, Regression, Logistic

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Truvada Plus Raltegravir
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes